CLINICAL TRIAL: NCT06703593
Title: Evaluation of the Impact of Alpha Lipoic Acid Administration on the Prevention of Doxorubicin-induced Cardiotoxicity in Breast Cancer Patients
Brief Title: Prevention of Doxorubicin-induced Cardiotoxicity in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British University In Egypt (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alaa jamal, Demonstrator and Teaching assistant at the Clinical Pharmacy Practice Department, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CL-2311
Record Dates: First submitted 2024-03-05; First posted 2024-11-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer Female
Keywords: Alpha lipoic acid, Anthracyclines induced Cardiotoxicity
MeSH Terms: interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alpha Lipoic acid intervention arm (Experimental): Alpha Lipoic acid 1200 mg daily for 6 months
  Interventions: Drug: Alpha lipoic acid
- No intervention arm (No Intervention): not taking Alpha Lipoic acid

INTERVENTIONS:
Drug: Alpha lipoic acid — ALA effectively inhibits nuclear factor-kappa B with subsequent decreasing proinflammatory cytokines production (TNF-α, IL-6) and increasing the release of anti- inflammatory cytokines such as interleukin-10 (Haghighatdoost and Hariri, 2019). Relying on the antioxidant and anti-inflammatory effect of Alpha lipoic acid confirmed by a variety of studies in vitro and in vivo, ALA is selected to be studied in Egyptian breast cancer patients who will be treated with doxorubicin including regimens.
  Other Names: Neuropatex; lipoic acid
  Arms: Alpha Lipoic acid intervention arm

SUMMARY:
According to the European Society of Cardiology 2022, the primary prevention of cancer therapyrelated cardiovascular toxicity during anthracycline chemotherapy include renin-angiotensin- aldosterone system blockers, beta-blockers, and mineralocorticoid receptor antagonists that have shown a significant benefit in preventing left ventricular ejection fraction (LVEF) reduction, but with no statistical differences in the incidence on the various other clinical outcomes as overt congestive heart failure (CHF). Also, other strategies have been investigated including; adjusting the infusion time and dose intensity of anthracyclines. Dexrazoxane and liposomal anthracyclines are currently approved in patients with high and very high chemotherapy-related cardiovascular disease (CTRCD) risk or who have already received high cumulative anthracyclines doses (Lyon, 2022). The incidence is about 4% when the dose of doxorubicin is 500-550 mg/m2, 18% when the dose is 551-600 mg/m2 and 36% when the dose exceeds 600 mg/m2 (Lefrak, 1973). Alpha-lipoic acid (ALA) was reported to have a cardioprotective role against doxorubicin-induced cardiotoxicity through attenuation of oxidative stress via scavenging reactive oxygen species (ROS), regenerating endogenous antioxidants including glutathione, vitamin E, and C, its metal chelation activity and its ability to repair oxidative damage. (Werida et al, 2022)

DETAILED DESCRIPTION:
ALA effectively inhibits nuclear factor-kappa B with subsequent decreasing pro- inflammatory cytokines production (TNF-α, IL-6) and increasing the release of anti- inflammatory cytokines such as interleukin-10 (FahimehHaghighatdoostabMitraHariri, 2019).

Relying on the antioxidant and anti-inflammatory effect of Alpha lipoic acid confirmed by a variety of studies in vitro and in vivo, ALA is selected to be studied in Egyptian breast cancer patients who will be treated with doxorubicin including regimens.

Aim of the study:

The aim of the current study is to evaluate the efficacy and tolerability of ALA administration and its impact on the occurrence of doxorubicin-induced cardiotoxicity in Egyptian women with breast cancer by evaluation of the following:

1. Evaluation of the occurrence of chemotherapy induced cardiotoxicity by;

   1. Changes in echocardiographic findings and serum levels of pro brain natriuretic peptide (pro-BNP) and cardiac troponins.
   2. Severity of DIC will be evaluated by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 For Heart Failure.
   3. Estimation of oxidative stress burden by measurement of MDA.
2. Evaluation of ALA safety by:

ALA safety will be monitored and assessed through patient face to face interviews (at the end of each cycle) and phone calls weekly about the occurrence of any of the following side effects: (Ex; insomnia, fatigue, diarrhea, and skin rash).

Patients will be followed up by monitoring of the side effect reporting card (intervention arm)

ELIGIBILITY:
Inclusion Criteria:

1. Women aged more than 18 years
2. Breast cancer diagnosis
3. Entering first cycle of chemotherapy containing ATC
4. Subject must be willing and able to sign an informed consent

Exclusion Criteria:

1. History of renal (serum creatinine greater than 2.0 mg/ml) or hepatic insufficiency (bilirubin> 3.0 mg/dl or serum albumin < 3.5 g/dl or prothrombin time < 60% in the absence of orally administered anticoagulant therapy or ultrasound signs of chronic liver damage
2. History of heart failure
3. Baseline LVEF < 50% determined by transthoracic echocardiogram
4. Current participation in any other clinical investigation
5. History of severe adverse reaction to Alpha lipoic acid
6. Concomitant use of Trastuzumab (HER2 positive patients)
7. Previous intake of alpha lipoic acid in the previous 3 months
8. Women with prior exposure to anthracyclines and neurotoxic agents (Cis-platin, vincristine, paclitaxel, docetaxel, foscarnet, isonicotinic acid hydrazide "INH,", etc.) in the last 6 months.
9. Presence of clinical evidence for severe cardiac illness (i.e., angina pectoris and arrhythmias)
10. Any condition that contraindicates chemotherapy (i.e., pregnancy, lactation)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 1. Women aged more than 18 years
  2. Breast cancer diagnosis
  3. Entering first cycle of chemotherapy containing ATC
  4. Subject must be willing and able to sign an informed consent
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in echocardiographic findings | Approximately few days ( less than a week ) before Cycle 1 "baseline" and after Cycle 4 "End Cycle" of Doxorubicin. Each cycle is 21 days.
  Elevation or maintenance of Ejection fraction percentage (EF %)
Changes in serum levels of pro brain natriuretic peptide (pro-BNP) and cardiac troponins | Just before Cycle 1 "baseline" and 1 hour after Cycle 4 "End Cycle" of Doxorubicin. Each cycle is 21 days.
  Decline in serum concentration of pro brain natriuretic peptide (pro-BNP) measured in picograms per milliliter (pg/mL) and cardiac troponins measured in picograms per milliliter (pg/mL).

SECONDARY OUTCOMES:
Changes in the oxidative stress marker malondialdehyde (MDA) | ust before Cycle 1 "baseline" and 1 hour after Cycle 4 "End Cycle" of Doxorubicin. Each cycle is 21 days.
  Decline in serum concentration of malondialdehyde (MDA) measured in micro mole / Litre

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, El-Sherouk City, Egypt

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication